CLINICAL TRIAL: NCT07077538
Title: A Single Center, Open, Prospective, Self-control Clinical Study on the Use of Amino Acid Peritoneal Dialysis Fluid in Diabetes Patients
Brief Title: Clinical Study of the Use of Amino Acid Peritoneal Dialysate in Diabetic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The People's Hospital of Gaozhou (Other)
Collaborators: Chengdu Qingshan Likang Pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, deng shanshan, Director, The People's Hospital of Gaozhou
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GYLLPJ-2025046
Record Dates: First submitted 2025-06-24; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Peritoneal Dialysis; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental)
  Interventions: Drug: Amino acid peritoneal dialysis solution

INTERVENTIONS:
Drug: Amino acid peritoneal dialysis solution — After breakfast daily, use a bag of amino acid (15) peritoneal dialysis solution (2L), followed by treatment with glucose peritoneal dialysis solution (lactate).

SUMMARY:
The study is a single center, open, prospective, self controlled clinical study. The patients with diabetes who are to be enrolled in peritoneal dialysis are to observe the changes of glycosylated hemoglobin relative to the baseline 90 days after using amino acid (15) peritoneal dialysis solution.

ELIGIBILITY:
Inclusion Criteria:

* Type I or II diabetes patients aged 18 to 75 years (including 18 and 75 years), regardless of gender;
* Stable peritoneal dialysis patients who have undergone peritoneal dialysis treatment for ≥ 3 months;
* Use 3-5 bags of peritoneal dialysis solution daily;
* 6.0%<glycated hemoglobin (HbA1c) level ≤ 8.5%;
* 90g/L ≤ Hemoglobin concentration ≤ 130g/L
* Stable use of erythropoietin and rosuvastatin;
* The fluctuation of carbohydrate energy supply ratio in the first 3 months before enrollment is less than 15%;
* Not using amino acid (15) peritoneal dialysis solution for the first 3 months before enrollment;
* Within the past month, the patient's prescription for hypoglycemic drugs has not been adjusted;
* Within the past month, the patient's dietary structure and food intake have remained stable.

Exclusion Criteria:

* Peritonitis has occurred within the past 3 months;
* Use Acodextrin peritoneal dialysis solution;
* Contraindications for the presence of amino acids (15) in peritoneal dialysis fluid:

  1. Individuals allergic to any component of amino acid (15) peritoneal dialysis fluid;
  2. Serum urea level>38 mmol/l;
  3. Metabolic acidosis (CO2 binding capacity<22mmol/L);
  4. Severe hypokalemia (blood potassium<2.5mmol/L);
  5. Various congenital amino acid metabolism abnormalities;
  6. Liver dysfunction (alanine aminotransferase levels exceeding 2.5 times the upper limit of normal);
* Combined hemoglobinopathies: such as thalassemia, sickle cell disease, etc;
* It is expected that kidney transplantation may be accepted during the trial period;
* Participated in other clinical studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To observe the changes of glycosylated hemoglobin (HbA1c) in peritoneal dialysis patients with diabetes after 90 days of using amino acid (15) peritoneal dialysis solution. | Day 0、Day 90

SECONDARY OUTCOMES:
To observe the changes of fasting blood glucose relative to the baseline after 30 and 90 days of using amino acid (15) peritoneal dialysate in diabetes patients undergoing peritoneal dialysis. | Day 0、Day 30、Day 90
To observe the changes of serum albumin relative to the baseline after 90 days of using amino acid (15) peritoneal dialysate in diabetes patients undergoing peritoneal dialysis. | Day 0、Day 90
To observe the changes of hemoglobin relative to the baseline after 90 days of using amino acid (15) peritoneal dialysate in diabetes patients undergoing peritoneal dialysis. | Day 0、Day 90
To observe the changes of prealbumin relative to baseline after 90 days of using amino acid (15) peritoneal dialysate in diabetes patients undergoing peritoneal dialysis. | Day 0、Day 90
To observe the relative baseline changes of daily urine volume and ultrafiltration volume after 30 and 90 days of using amino acid (15) peritoneal dialysate in diabetes patients undergoing peritoneal dialysis. | Day 0、Day 30、Day 90
To observe the changes of Kt/v in peritoneal dialysis patients with diabetes 90 days after using amino acid (15) peritoneal dialysis solution. | Day 0、Day 90
To observe the changes of Ccr in peritoneal dialysis patients with diabetes 90 days after using amino acid (15) peritoneal dialysis solution. | Day 0、Day 90
To observe the changes of hypoglycemic drugs in peritoneal dialysis patients with diabetes 90 days after using amino acid (15) peritoneal dialysis solution. | Day 0、Day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Ethics Committee of Gaozhou People's Hospital, Gaozhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duong U, Mehrotra R, Molnar MZ, Noori N, Kovesdy CP, Nissenson AR, Kalantar-Zadeh K. Glycemic control and survival in peritoneal dialysis patients with diabetes mellitus. Clin J Am Soc Nephrol. 2011 May;6(5):1041-8. doi: 10.2215/CJN.08921010. Epub 2011 Apr 21. PMID 21511838
- [Background] Qayyum A, Chowdhury TA, Oei EL, Fan SL. Use of Continuous Glucose Monitoring in Patients with Diabetes Mellitus on Peritoneal Dialysis: Correlation with Glycated Hemoglobin and Detection of High Incidence of Unaware Hypoglycemia. Blood Purif. 2016;41(1-3):18-24. doi: 10.1159/000439242. Epub 2015 Oct 20. PMID 26960210
- [Background] Gomez AM, Vallejo S, Ardila F, Munoz OM, Ruiz AJ, Sanabria M, Bunch A, Morros E, Kattah L, Garcia-Jaramillo M, Leon-Vargas F. Impact of a Basal-Bolus Insulin Regimen on Metabolic Control and Risk of Hypoglycemia in Patients With Diabetes Undergoing Peritoneal Dialysis. J Diabetes Sci Technol. 2018 Jan;12(1):129-135. doi: 10.1177/1932296817730376. Epub 2017 Sep 20. PMID 28927285